CLINICAL TRIAL: NCT02023411
Title: To Study the Efficacy of Teriparatide in Improving Remodeling of Foot Bones in Chronic Charcot Neuroarthropathy in Patients With Diabetes Mellitus.
Brief Title: Efficacy of Teriparatide in Diabetic Inactive Charcot Neuroarthropathy of Foot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Asst Professor , Department of Endocrinology, Post graduate institute of medical education and research, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABAR-1072013
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Neuropathic Arthropathy
Keywords: Teriparatide; Inactive Charcot's neuroarthropathy
MeSH Terms: interventions — Teriparatide; Parathyroid Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- teriparatide (Active Comparator): 10 diabetic patients with inactive Charcot's foot who are calcium and Vit.D sufficient will receive 20 microgram of teriparatide , subcutaneous between 8-9 p.m., daily.
  Interventions: Drug: Teriparatide
- placebo (Placebo Comparator): 10 diabetic patients with inactive Charcot's foot who are calcium and Vit.D sufficient will receive placebo , subcutaneous between 8-9 p.m. , daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Teriparatide — recombinant human parathyroid hormone (1-34) subcutaneous every day at 8-9 pm
  Other Names: parathyroid hormone; recombinant human parathyroid hormone
  Arms: teriparatide
Other: Placebo — Placebo
  Arms: placebo

SUMMARY:
Diabetic foot represents a major medical , social and economic problem worldwide.

Charcot's neuroarthropathy, being a common cause of diabetic foot, has been an intriguing topic of research for endocrinologists, podiatrists and surgeons. After its first description by JEAN-MARTIN CHARCOT in 1868, many theories have been put forward regarding its pathophysiology , but not much research has been done for its prevention and treatment , specially the inactive stage.

The course of Charcot 's neuroarthropathy is triphasic , with the diagnosis being usually missed in the active stage, henceforth the patients often come to us with a deformed foot. As a consequence , the osteoclastic activity in active stage renders the foot bones demineralized and weak, thus being susceptible to fracture and fragmentation.

Teriparatide is recombinant human (1-34) parathyroid molecule that has been approved for post-menopausal osteoporosis and in men with primary or secondary osteoporosis. It acts by preferentially stimulating osteoblast over osteoclast activity resulting in new bone formation and an increase in the rate of bone remodeling which manifest as an increase in skeletal mass and bone mineral density .

Keeping the pathophysiology of Charcot's foot in mind, teriparatide may be used as potential treatment for inactive Charcot's neuroarthropathy but there are no studies or randomized trials in this setting, till date. We hypothesize that teriparatide may increase the remodeling of foot bones in Charcot's neuroarthropathy, improve bone mineral density, subsequently leading to a reduction in the risk of fractures and progression of deformities. This study plans to compare the effects of teriparatide in diabetes patients with inactive Charcot's foot in a placebo controlled design.

DETAILED DESCRIPTION:
Charcot neuroarthropathy (CN) was first described by Jean-Martin Charcot in a patient with tabes dorsalis who recognized that peripheral neuropathy could lead to neuropathic joints. This condition has many names, including Charcot osteoarthropathy, neuropathic osteo- arthropathy, and many others. Charcot foot may occur as a complication of neurosyphilis, syringomyelia, leprosy, poliomyelitis, congenital neuropathy and diabetes mellitus , the latter currently being the most common cause of CN. Since the description of CN in 1883, its pathophysiology remains an enigma, and there are no strict guidelines for the treatment of this disorder.

India has more people living with diabetes than any other country of the world and diabetic foot is one of the common diabetic complications found in India. The prevalence of Charcot foot in diabetes is not clearly known (0.1% to nearly 30%), but it is now appreciated that the condition is not as infrequent as might be generally thought. CN is characterized by progressive destruction of bones and joints of the foot with accompanying osteopenia. The current belief is that once the disease is triggered in a susceptible individual, it is mediated through a process of uncontrolled inﬂammation in the foot. This inﬂammation leads to osteolysis and is indirectly responsible for the progressive fracture and dislocation that characterizes its presentation.

The pathophysiologic event is cytokine- driven elevation of the receptor activator of nuclear factor kappa B ligand (RANKL), which, in turn, enhances the synthesis of nuclear factor kB (NF-kB). The latter promotes osteoclast maturation and osteoclastic activity, leading to osteoporosis in the affected bones. In parallel , NF-kB enhances the production of osteoprotegerin from osteoblasts, in order to provide an antagonist of RANKL and mitigate its effects. Ultimately, the cascade of all pathophysiologic changes leads to the development of the Charcot's foot and demineralization of bones.

If the condition is correctly diagnosed and the patient is appropriately immobilized, the local inflammation will subside and further bony destruction including progressive loss of mineral density may be prevented. But the diagnosis of CN is frequently missed in the active phase in almost 25% of cases. In the inactive stage, signs of local inﬂammation progressively recede, redness subsides, and the difference in skin temperature between the two feet diminishes. Most of the patients coming to our diabetes clinic present in the inactive phase with stable foot deformities viz rocker bottom deformity, loss of longitudinal or transverse arches, bony prominence (medial convexity) and significant demineralization of bones. These foot deformities result in abnormal high-pressure areas that are particularly prone to ulceration; a consequence of continued weight bearing.

Recombinant human parathyroid hormone fragment (teriparatide) is an anabolic therapy , that preferentially stimulates osteoblast over osteoclast activity resulting in new bone formation and an increase in the rate of bone remodeling. These effects manifest as an increase in skeletal mass, bone mineral density (BMD) and bone strength, subsequently leading to a reduction in the risk of fractures. It has been well established that teriparatide increases bone remodeling in the skeleton through histomorphometry studies and measurements of bone turnover markers (BTM), and recently direct measurements of the effect of teriparatide on the site-specific metabolic activity of the skeleton has been shown in patients of osteoporosis.

Radionuclide bone scan imaging using the radiopharmaceutical 99Technetium-methylene diphosphonate (MDP) has a useful role in both clinical practice and research to investigate metabolic bone diseases and response to treatment. In clinical practice, bone scans are reported solely on a qualitative visual interpretation of images allowing for the detection of discrete changes in the skeleton in areas of focal tracer uptake. An increased 99mTc-MDP skeletal uptake with teriparatide is seen in patients with osteoporosis indicating an increased bone formation which was supported by BTM increases. Recently, quantitative bone scintigraphy with MDP is described as a more sensitive tool to study the bone-remodeling process even in CN. The potential utility of quantitative bone scanning for the diagnosis and more importantly for CN activity is suggested. However, translating visual assessments into quantitative data with F18 PET/ SPECT CT to study the regions of interest (ROI) and assess the response to teriparatide will be more specific.

The role of teriparatide in diabetes patients with CN has not been studied, till date. Keeping the pathophysiology of CN in mind, the present study plans to assess the efficacy of teriparatide in chronic CN by studying the change in bone remodeling as quantitated by F18 SPECT CT, BMD and markers of bone turnover. We will also assess the benefits of teriparatide, if any, on the foot morbidity i.e incidence of fractures, progression of deformity or need for amputation over the follow up period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical criteria:

   1. No warmth or redness of foot.
   2. Difference in temperature between two foot < 2 degree Centigrade.
   3. If deformity present , patient able to walk without aid.
   4. History of resolved active Charcot's neuroarthropathy of foot.
2. Radiological criteria: Plain X-ray foot (weight bearing lateral and oblique) showing at least 3 of the following features -

   1. Foot deformity.
   2. Joint subluxations/dislocations.
   3. Smoothening /Rounding of bone fragments.
   4. Subchondral sclerosis/erosions.
   5. Callus formation.
   6. Joint space collapse.

Exclusion Criteria:

1. Active inflammatory phase of Charcot's neuroarthropathy.
2. Active on inactive Charcot's neuroarthropathy.
3. Osteomyelitis of foot bones.
4. Peripheral vascular disease.
5. Osteoporosis (T score less than or equal to -2.5 at lumbar spine or hip).
6. Renal failure ( estimated Glomerular Filtration Rate < 60 ml/min).
7. Previous/present bone malignancy.
8. Previous malignancy with metastases to bone.
9. Received teriparatide earlier.
10. Hyperparathyroidism.
11. Paget's disease of bone.
12. Pregnant women.
13. Received bisphosphonates in previous 18 months.
14. Patients with ulcer on the involved foot.
15. Patients previously taking Pioglitazone. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, DM, Principal Investigator — PGIMER, Chandigarh
Locations (2):
- India (2):
  - Deptt of Endocrinology, Chandigarh
  - PGIMER, Chandigarh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment performed from January 2016 and closed on December 2017
Groups:
- Teriparatide: Intervention Arm
- Placebo: Normal saline will be subcutaneously administered at 8 pm daily
Period: Overall Study
Arm/Group | Teriparatide | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Each Participant Foot was considered as one unit. Only one foot of each participant was included.
Groups:
- Intervention Arm: Teriparatide 20 microgram administered Subcutanoeous daily
- Placebo: Normal saline administered Subcutanoeous daily
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 52.3 (8.8) | 55 (7.8) | 53.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 10 | 10 | 20
SUVmax of affected foot [Median (Inter-Quartile Range); unit: g/ml] — F18 PETCT of affected foot was performed at baseline and SUV max ta the affected area of the foot was recorded
  g/ml | 27.6 [20.8 to 45.1] | 27.2 [15.3 to 38.5] | 27.4 [18.1 to 41.2]

OUTCOME MEASURES:

1. Primary Outcome: SUV Max on PET/CT Scan at 12 Months
Description: F18 PET/CT scan of foot was performed at baseline and at 12 months following intervention. Main outcome measure was Standardised Uptake value (SUV max) with intervention. A higher score on the scale suggest better outcome
Time Frame: 12 months
Population: intervention versus placebo
Measure: Mean (Standard Deviation); unit: g/ml
Groups:
- Placebo: Normal saline subcutaneous injection
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 10 | 10
g/ml | 26.1 (11.4) | 22.9 (10.4)

2. Secondary Outcome: Clinical Events
Description: Any of the following will be taken as a secondary end point:
  The number of participants with
  1. new onset fracture
  2. new onset/progression of deformity
  3. amputation
Time Frame: 12 months
Population: Participants receiving TEriparatide were observed for secondary outcomes of fractures, deformities and amputation
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo normal saline was given
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: Intervention is not known to be associated with mortality
Groups:
- Teriparatide: 10 diabetic patients with inactive Charcot's foot who are calcium and Vit.D sufficient will receive 20 microgram of teriparatide , subcutaneously between 8-9 p.m., daily.
  Teriparatide: recombinant human parathyroid hormone (1-34) subcutaneously every day at 8-9 pm
- Placebo: 10 diabetic patients with inactive Charcot's foot who are calcium and Vit.D sufficient will receive placebo , subcutaneously between 8-9 p.m. , daily.
  Placebo: Placebo
Arm/Group | Teriparatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teriparatide (N=10) | Placebo (N=10)
Hypercalcemia (Endocrine disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Small sample size Shorter follow-up duration of 12 months. Arbitrary value for SUVmax of ≥2.5 as a significant value No Histomorphometric analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT02023411/Prot_SAP_000.pdf